CLINICAL TRIAL: NCT03793595
Title: Oxygen Consumption and Heart Rate Response to Battle Rope Exercise Protocol Versus Upper Extremity Arm Bike Test in Adults With Spinal Cord Injury
Brief Title: O2 Consumption and Heart Rate Response to Battle Rope Exercise Protocol Versus UE Arm Bike Test in Adults With SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Wayne Brewer, Associate Professor, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2019-34
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Spinal Cord Injury at T2 and Below

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Seated Battle Ropes Protocol (Experimental)
  Interventions: Device: Seated Battle Ropes Protocol
- Seated Upper Extremity Arm Bike (Active Comparator)
  Interventions: Device: Seated Upper Extremity Arm Bike

INTERVENTIONS:
Device: Seated Battle Ropes Protocol — Participants will begin swinging the rope as previously described in the seated position using the double arm swing technique for 15 seconds at a cadence of 100 beats/ minutes with a 45 second rest break repeated 10 times.
  Arms: Seated Battle Ropes Protocol
Device: Seated Upper Extremity Arm Bike — A modified Young Men's Christian Association (YMCA) cycle test will be performed.
  Arms: Seated Upper Extremity Arm Bike

SUMMARY:
The purpose of this study is to compare energy expenditure and metabolic outcomes of a novel seated battle rope protocol to seated maximal ramped upper extremity ergometry protocol in subjects with spinal cord injury.

DETAILED DESCRIPTION:
1. Subjects will be scheduled for the first testing session after informed consent is obtained.
2. Subjects will fill out PAR-Q+ to determine readiness for exercise testing
3. Subjects will fill out additional Questionnaire to determine exclusion based on medical history
4. Prior to the physical performance tests, each participant will be fitted with a mask that covers their face. This mask will be attached to a portable metabolic analyzer (Cosmed k5b). This device collects the air expired which allows for energy expenditure to be estimated.
5. Each participant will be fitted with the proper sized mask that is connected to a small computer and power source supported at their upper back.
6. A polar heart rate strap monitor will be worn around the chest. As the participant performs the physical performance tests, the Cosmed K5b measures the amount of carbon dioxide and oxygen from each breath to estimate the amount of energy expended during this task.

Session one:

1. Prior to beginning the testing, testing procedure will be explained to participants
2. Subjects blood pressure will be measured, and if a subject's average systolic or diastolic blood pressure exceeds 140 or 90 mmHg, respectively, the subject will be asked to return another day to perform the study procedures. If the blood pressure remains elevated on either one of these measures, the subject will be excused from this study.
3. Subjects will then perform either the upper extremity cycling protocol or battle ropes protocol first. The other will be performed on the subsequent testing date
4. If the subject is performing the upper extremity arm cycle test:

   Each subject will perform a modified version of the ramped YMCA cycle test using a Upper Extremity Cycle Ergometer and a portable metabolic cart
   * The ramped version of the YMCA cycle test will begin with the subject cycling at a workload of 25 watts at a rate of 60 revolutions per minute (rpm) using a metronome set at 120 beats per minute.
   * Each subject will pedal for 3-minute warm-up period at the 10 watts with the 60 rpm rate. After the 3-minute warm-up, the workload will increase by 10 watts each minute starting at 25 watts at pedal rate of 60 rpm until the subjects meets the termination criteria as described below.
5. The portable metabolic cart is an instrument that measures levels of expired gases from the subject as he or she exercises that will be analyzed and displayed on a computer monitor. The subject will wear a face mask during the test. A Polar® heart rate monitor will be worn on the chest, directly on the skin of each subject to obtain heart rate measurements.
6. The goal is for the participant to perform the ramped exercise test using the protocol described above and below until one or more of the following occurs, at which time the test will be terminated: the participant requests the test to be stopped, a respiratory exchange ratio of >1.0 is achieved, or one of the following physiologic and/or subjective signs/symptoms are present:

   * i. A drop in systolic blood pressure >10 mmHg with the increasing work load
   * ii.An increase in systolic and/or diastolic blood pressure >250 mmHg or 115 mmHg, respectively.
   * iii.Reported chest or arm pain (angina)
   * iv.Severe shortness of breath, cyanosis, pallor, lightheadedness, dizziness or confusion
   * v.No increase in heart rate despite increase in work load
   * vi.Complaints of severe fatigue
   * vii.The subject is unable to maintain a pedal rate of 50 rpm
   * viii.Borg 6-20 Perceived exertion scale score >=20
7. The subjects heart rate will be recorded at the last 15-30 seconds of each minute during the test.
8. Each subject's blood pressure will be taken before the test commences, every three minutes during the test and once the test procedure is terminated.
9. The Borg 6-20 perceived exertion scale will be used to monitor the participant's rating of perceived exertion every three minutes during the test. If at any time during the test, the subject rates his or her perceived level of exertion at a level of 20, the test will be terminated.
10. Session two: will occur at least three days after session one.
11. If the subject is performing the sitting battling rope:

    * a. A 10 to 15-minute demonstration will be provided to each subject on the proper use of the battling ropes using the double arm swing technique
    * b. A 30 foot,1.5-inch diameter rope that will be anchored to a large weight

      c. Each subject will position him/herself in their manual wheelchair with feet flat on the floor or foot rests at shoulder width apart.
    * d. The subject's manual wheelchair will be secured using dumbbells and weights as pictured below
    * e. A 3-minute warm up period will be given to each subject prior to the exercise protocol

      f. The subject will be fitted with a face mask attached to the metabolic cart as described previously.

      g. On command, each subject will begin swinging the rope as previously described in the seated position using the double arm swing technique for 15 seconds at a cadence of 100 beats/ minutes with a 45 second rest break repeated 10 times.

      h. At each rest break, the subject will be asked to rate his/her levels of exertion using the Borg 6-20 as described previously.
    * i. If a subject cannot complete the double arm rope swing at the required cadence or if the rope does not undulate through the entire length of the rope towards the anchor point, or if the subject requests to stop, the protocol will be terminated.
12. Reusable Mask cleaning procedure, performed following each participant

    * a. the following parts must be 1) rinsed with warm soapy water, 2) soaked in CITADEX solution 15 minutes, 3) rinsed with cool running water again, 4) laid out to dry:
    * b. Turbine (fan tube)
    * c. Flowmeter seal (black plastic cone ring)
    * d. Flowmeter cap (tan circle with black and silver emblem on it)
    * e. Face mask (blue plastic inserted vertically to avoid air pockets on interior)
13. After each use, the following parts must be wiped down with baby wipes and at the end of the day must be soaked in soapy water for 10 minutes then wrung out and laid out to dry:

    * a. Head strap
    * b. Polar monitor strap
    * c. After each use, the following must be wiped with a disinfectant wipe:
    * d. Polar hear monitor

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord lesion T2 or below
* Individuals with spinal cord injury for greater than six months
* Utilize manual wheelchair for greater than 10 hours a day

Exclusion Criteria:

* Current complaints of spinal, lower extremity or upper extremity pain or musculoskeletal disorder that prevents the subject from performing repetitive upper extremity cycling or grasping and swinging the weighted ropes against the floor
* A current diagnosis of a chronic or acute cardiovascular, metabolic, renal or pulmonary disease including use of a pacemaker
* Anyone currently taking beta blocker medication
* Anyone with blood pressure >140/90 at the time of testing or with in the 2 weeks prior to testing
* Diagnosed sickle cell disease or sickle cell trait
* Severe spasticity or joint contracture preventing subject from performing upper extremity cycling or swinging of weighted ropes
* Subjects with current decubital ulcers
* History of autonomic dysreflexia in the last 6 months
* Require physician follow-up prior to starting exercise based on PAR-Q+ questionnaire

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness as assessed by maximum oxygen uptake (VO2max) | about 10-15 minutes after start of the protocol
  VO2max will be measured using a portable metabolic cart (Cosmed k5b).

SECONDARY OUTCOMES:
Heart Rate | about 10-15 minutes after start of the protocol
Rate of perceived exertion as assessed by the Borg 6-20 Perceived exertion scale | about 10-15 minutes after start of the protocol
  The Borg 6-20 Perceived exertion scale score ranges from 6-20, higher score indicates a worse outcome.
Blood pressure | about 10-15 minutes after start of the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Wayne A Brewer, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No